CLINICAL TRIAL: NCT00809380
Title: Parental Presence During Fracture Reduction in Children at the Emergency Department; A Randomized Controlled Trial
Acronym: PP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study ws terminated because of a too low recruitment rate.
Sponsor: St. Justine's Hospital (Other)
Collaborators: Association des Médecins d'Urgence du Quebec (Unknown)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, MSc, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PP
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Conscious Sedation; Anxiety
Keywords: Conscious sedation; Parental presence; Invasive procedure; Children; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parental presence (Experimental): Patients in the study group will be accompanied by one of their parents for the whole procedure. Before this, a short explanation of the procedure, the patient's expected behavior during the procedure and what roles parents should play will be given to the parent by the research assistant. Parents will be seated close to the patient's head and will wear radiology proof gowns. If deemed necessary by the attending physician or if their behavior becomes unacceptable, parents can be asked to leave the procedure room at any given time. Parents will be allowed to leave the procedure room if they wish to at any time during the procedure.
  Interventions: Behavioral: Parental presence
- Control (Active Comparator): One parent will stay with their child until he is in the procedure room and conscious sedation has begun. He will then be asked to leave the room and wait in an adjoining waiting room. The attending physician will invite the parent back in the room once the reduction is complete and the cast is done.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Parental presence — Patients in the study group will be accompanied by one of their parents for the whole procedure. Before this, a short explanation of the procedure, the patient's expected behavior during the procedure and what roles parents should play will be given to the parent by the research assistant. Parents will be seated close to the patient's head and will wear radiology proof gowns. If deemed necessary by the attending physician or if their behavior becomes unacceptable, parents can be asked to leave the procedure room at any given time. Parents will be allowed to leave the procedure room if they wish to at any time during the procedure.
  Arms: Parental presence
Behavioral: Control — One parent will stay with their child until he is in the procedure room and conscious sedation has begun. He will then be asked to leave the room and wait in an adjoining waiting room. The attending physician will invite the parent back in the room once the reduction is complete and the cast is done.
  Arms: Control

SUMMARY:
Though much attention has been given to the practice of parental presence during invasive procedures in children in the ED, few studies have examined the patient's perspective. The only study to have addressed this issue used a single visual analog scale, which is not a well validated tool to assess children's distress level. Furthermore, no studies have assessed parental presence during fracture reduction; only a few incidental cases were reported in the literature. Finally, most studies evaluating parental presence had methodological limitations because of the absence of a control group.

The investigators seek to assess whether parental presence during fracture reduction under sedation, in children 8 to 18 years of age, decreases anxiety levels in both parents and children.

ELIGIBILITY:
Inclusion criteria for patients:

* Patients aged 8 to 18 years old.
* Patients requiring fracture reduction under conscious sedation by emergency department attending physician.
* Patients able to understand basic spoken English or French.

Inclusion criteria for parents:

* Parents able to understand basic spoken English or French.

Exclusion criteria for patients:

* Patients with moderate to severe mental retardation
* Patients with altered mental status or intoxication
* Patients with hemodynamic instability or several traumatic injuries (other than fractures) - these patients require several treatments and may not have time to complete our study.

Exclusion criteria for parents:

* Parents presenting unacceptable behaviors for family presence

  * Uncooperative
  * Physically aggressive, combative
  * Threatening and argumentative
  * Unstable emotionally or cannot be calmed
  * Intoxicated or altered mental status
  * Suspicion of child abuse
  * Suspected perpetrator of violent crime
* Parents with moderate to severe mental retardation.
* Pregnant parent

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The children's anxiety will be measured using the State-Trait Anxiety Inventory (STAI) score (in children older than 12) or State-Trait Anxiety Inventory for children (STAIC) scores (in children from 8 to 12 years old) | at discharge (2 hours post randomisation)
The parents' anxiety will be measured using the STAI scores. | At discharge (approximately 2 hours post randomisation)

SECONDARY OUTCOMES:
Procedure time | 1 hours
Doses and types of medications used | 1 hour
Fracture reduction success and failure rates | 1 hour
Attempt of reduction by the residents | 1 hour
STAI and STAIC scores in children at induction of conscious sedation will be compared between both groups | 1 hour
Children's anxiety levels will also be assessed with the modified Yale Preoperative Anxiety Scale | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, Principal Investigator — St. Justine's Hospital; Nathalie Gaucher, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada